CLINICAL TRIAL: NCT00676260
Title: Effect of Pioglitazone 15 mg or 30 mg on Microcirculation in Type 2 Diabetes Patients Treated With Insulin
Brief Title: Efficacy of Pioglitazone on Microcirculation in Type 2 Diabetes Patients Treated With Insulin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD4833/EC412; U1111-1114-1082 (Registry Identifier: WHO)
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pioglitazone QD (Experimental)
  Interventions: Drug: Pioglitazone
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 15 mg to 30 mg, tablets, orally, once daily for up to 10 weeks
  Other Names: Actos; AD4833
  Arms: Pioglitazone QD
Drug: Placebo — Pioglitazone placebo-matching tablets, orally, once daily for up to 10 weeks
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to measure microcirculation in type 2 diabetes patients with peripheral edema who are taking pioglitazone, once daily (QD).

DETAILED DESCRIPTION:
Pioglitazone is a thiazolidinedione compound with a mode of action as a peroxisome proliferator-activated receptor gamma agonist. Activation of this receptor causes increased transcriptional activity at a number of locations that are important to carbohydrate and lipid (fat) metabolism. Insulin resistance is reversed by enhancing the action of insulin, thereby promoting glucose utilization in peripheral tissues, suppressing gluconeogenesis in the liver, and reducing lipolysis at the adipocyte.

In previous studies of pioglitazone, peripheral edema (swelling in the hands, feet, and legs) was reported as an adverse event more often in pioglitazone groups and appears to be a dose dependent phenomenon with pioglitazone. The incidence of peripheral edema in monotherapy studies was 3.2% in pioglitazone patients compared with 0.7% placebo patients and was reported more by females than males. This incidence was higher when pioglitazone was combined with sulphonylurea or insulin (5.9% and 15.6%, respectively). In comparison, the incidence of edema, when sulphonylurea or insulin was combined with placebo, was 2.1% and 7.5%, respectively.

This study is designed to identify the mechanisms underlying peripheral edema formation with pioglitazone in patients with Type 2 diabetes.

Individuals who participate in this study will provide written informed consent and will be required to commit to a screening visit and approximately 4 additional visits at the study center. Study participation is anticipated to be about 10 to 12 weeks (or approximately 3 months). Multiple procedures will occur at each visit which may include fasting, blood collection, urine collection, physical examinations and electrocardiograms.

ELIGIBILITY:
Inclusion Criteria:

* Stable glycemic control glycosylated hemoglobin between 6.5 and 10%) in the two months prior to the study.
* Type 2 diabetes treated by diet and stable dose of insulin (alone or with metformin) in the three months prior to the study.
* Female patients must have been postmenopausal, had a hysterectomy, or were surgically sterilized.

Exclusion Criteria:

* Has Type 1 diabetes.
* Has an episode of hypoglycemia requiring medical assistance three months prior to the study.
* Has peripheral artery disease (including Raynaud's syndrome) confirmed by an Ankle Brachial Pressure Index less than 0.9.
* Has severe chronic venous insufficiency as evidenced by venous ulceration or subcutaneous serum deposits.
* Has vascular autoimmune disease, had received a renal transplant, or were receiving dialysis.
* Has had heart failure (New York Heart Association I to IV), left ventricular hypertrophy evident from the ECG, or myocardial infarction 12 months prior to start of study.
* Has Subject had uncontrolled hypertension or familial polyposis coli.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Non steroidal anti-inflammatory Drugs (except for aspirin at anti-aggregant doses), oral anti-diabetic drugs (except metformin), calcium-channel blockers, and diuretics at anti-edema doses are excluded from the study.
  * Treatment with systemic corticosteroids within four weeks prior to enrolment and during the study was not allowed.
  * Patients who have taken beta-blockers are to have been on a stable dose for four weeks before entry in the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2002-12; Primary Completion 2004-08 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Capillary filtration capacity. | Final Visit

SECONDARY OUTCOMES:
Isovolumetric venous pressure. | Final Visit
Capillary pressure. | Final Visit
Postural vasoconstriction. | Final Visit
Maximum blood flow. | Final Visit
Capillary recruitment. | Final Visit
24-hour ambulatory blood pressure. | Final Visit
Interleukin-6 | Final Visit
C-Reactive Protein. | Final Visit
Vascular Endothelium Growth Factor. | Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Exeter, United Kingdom

REFERENCES:
- [Result] Tooke JE, Elston LM, Gooding KM, Ball CI, Mawson DM, Piper J, Sriraman R, Urquhart R, Shore AC. The insulin sensitiser pioglitazone does not influence skin microcirculatory function in patients with type 2 diabetes treated with insulin. Diabetologia. 2006 May;49(5):1064-70. doi: 10.1007/s00125-006-0168-9. Epub 2006 Mar 1. PMID 16508777
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI